CLINICAL TRIAL: NCT06915233
Title: A Prospective, Open-label, Randomized, Concurrent Active-controlled, Longitudinal, Multicenter, Phase 3 Clinical Study of the Safety and Efficacy of MACI in Patients With Symptomatic Chondral or Osteochondral Lesions of the Talus (MASCOT)
Brief Title: A Study of MACI in Patients Aged 17 to 65 Years With Symptomatic Chondral or Osteochondral Defects of the Ankle
Acronym: MASCOT
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Vericel Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 55-2410-01
Record Dates: First submitted 2025-04-01; First posted 2025-04-08 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Chondral Defect; Articular Cartilage Defect
Keywords: Bone Diseases; Musculoskeletal Diseases; Connective Tissue Diseases; Osteochondritis; Cartilage Diseases
MeSH Terms: conditions — Bone Diseases; Musculoskeletal Diseases; Connective Tissue Diseases; Osteochondritis; Cartilage Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MACI (Experimental): autologous cultured chondrocytes on porcine collagen membrane
  Interventions: Biological: autologous cultured chondrocytes on porcine collagen membrane
- Bone Marrow Stimulation (Active Comparator): Surgical procedure
  Interventions: Procedure: Bone Marrow Stimulation

INTERVENTIONS:
Biological: autologous cultured chondrocytes on porcine collagen membrane — An autologous cellularized scaffold product being studied for the repair of symptomatic, single or multiple full-thickness cartilage defects of the talus with or without bone involvement in adults.
  Arms: MACI
Procedure: Bone Marrow Stimulation — A surgical awl or microdrill will be used to make multiple holes in the exposed base of the lesion. The microfracture procedure should result in holes that are approximately 3 to 4 mm apart.
  When fat droplets can be seen coming from the marrow cavity, the appropriate depth (approximately 2 to 4 mm) has been reached.
  The released marrow elements (including mesenchymal stem cells, growth factors, and other healing proteins) form a surgically induced clot that provides an enriched environment for new tissue formation.
  Arms: Bone Marrow Stimulation

SUMMARY:
The objective of this study is to demonstrate the superiority of MACI (autologous cultured chondrocytes on porcine collagen membrane) versus Bone Marrow Stimulation in the treatment of patients aged 17 to 65 years with symptomatic articular chondral or osteochondral defects of the talus.

DETAILED DESCRIPTION:
This is a 2-year prospective, multicenter, two-arm, parallel-group open-label clinical trial in which a total of 309 subjects, ages 17 to 65, will be randomized 2:1 to receive a 1-time treatment in the ankle with MACI or arthroscopic BMS.

After meeting screening criteria at the initial visit (Visit 1), all subjects will have an index ankle arthroscopy within 8 weeks to further assess study eligibility. During the index ankle arthroscopy (Visit 2), patients will be further evaluated against entry criteria. Cartilage lesion size will be measured before any cartilage repair procedure and randomization. Only subjects with at least 1 lesion ≥ 1.2 cm² on the talus will be eligible for inclusion in the study.

All subjects who meet the eligibility criteria and are considered suitable for treatment in the study by their surgeon will have a cartilage biopsy taken prior to randomization to study treatment. Eligible subjects will be randomized 2:1 to receive either MACI or Bone Barrow Stimulation. Subjects randomized to Bone Marrow Stimulation will undergo the procedure during the Visit 2 ankle arthroscopy. Subjects will be asked to follow a recommended postoperative rehabilitation program.

All biopsied tissue will be sent to the Vericel Corporation manufacturing facility in Massachusetts, where the sample will be processed to isolate the autologous chondrocytes, undergo cell culture expansion through at least the primary phase, and cryopreservation. Additional expansion of the cells will occur after the MACI implantation surgery has been scheduled.

Subjects assigned to the MACI treatment arm will return within 5-12 weeks of the Visit 2 ankle arthroscopy to undergo MACI implantation procedure via arthrotomy (Visit 3). Subjects will be asked to follow a recommended postoperative rehabilitation program.

All subjects will be assessed post-study treatment at Weeks 6 and 12 for safety and at Weeks 24, 36, 52, 78, and 104 for safety and efficacy. Rehabilitation status will be monitored at all post-treatment visits until considered complete.

ELIGIBILITY:
Inclusion Criteria:

1. Age 17 to 65 at the time of planned randomization visit (Visit 2).
2. One or more symptomatic chondral or osteochondral lesion/s as defined by FAOS Pain score ≤ 50 and FAOS Function (SRA) score ≤ 50.
3. International Cartilage Repair Society (ICRS) Score Grade 3 or 4 chondral or osteochondral lesion/s located on the talus with or without cysts, including shoulder lesions (lesions on the talar neck), and amenable to treatment with the surgical procedure specified at randomization.
4. At least 1 lesion ≥ 1.2 cm².
5. Written informed consent and assent (as applicable) per Institutional Review Board (IRB) requirements.
6. Subject will refrain from using Non-steroidal Anti-inflammatory Drugs (NSAIDS) for 12 weeks post-study treatment. (Post-surgical use of low-dose aspirin for clot prevention is acceptable).
7. Subject will restrict pain medication to over-the-counter analgesics (NSAIDs or acetaminophen/paracetamol) after 12 weeks post-study treatment.
8. Subject must have Hematocrit ≥30.0%; White Blood Cell count ≤14,000 cells/μL; Platelet Count ≥50,000 platelets/μL; Creatinine ≤2.0 mg/dL; and International Normalized Ratio (INR) ≤1.6.

Exclusion Criteria:

1. Lesions with an underlying bony defect depth of > 5 mm.
2. Any surgery on the target joint within 24 weeks prior to Visit 1 (not including diagnostic ankle arthroscopy).
3. Previous investigational drug, biologic or device use within 12 weeks prior to Visit.
4. Avascular necrosis of the target ankle.
5. Symptomatic musculoskeletal conditions in the lower limbs that could impede measurement of efficacy for the target ankle joint.
6. Subjects with "kissing lesions" (bipolar lesions, involving both the tibia and talus), or with bilateral lesions in both ankles.
7. Subjects with lesions that require an osteotomy procedure to allow for MACI implantation as determined at the time of ankle arthroscopy (Visit 2).
8. Concomitant systemic inflammatory diseases or other conditions that affect the joints (e.g., rheumatoid arthritis, metabolic bone disease, psoriasis, symptomatic chondrocalcinosis).
9. History of advanced or severe osteoarthritis of the ankle as determined by prior surgical history confirming no joint space (i.e., "bone on bone") or radiographic evidence of Modified Kellgren-Lawrence Grade 4 arthritis (i.e., osteophytes on lateral and medial malleoli and at the tibiotalar joint margins, narrowing of the joint space width > 50%, and tibiotalar sclerosis), Van Dijk Grade III (i.e., total or subtotal destruction of the joint space) or the equivalent.
10. Known history of septic arthritis in the target ankle joint within 1 year prior to Visit 1.
11. Current malignancy or treatment for malignancy within the past 5 years prior to Visit 1, excluding non-melanoma skin cancer.
12. Known history of hypersensitivity to gentamicin, other aminoglycosides, or products of porcine or bovine origin.
13. Females who are pregnant or lactating.
14. Patients who, in the opinion of the Investigator, have significant medical or psychosocial problems that warrant exclusion. Examples of significant problems included but are not limited to:

    1. Any condition that has potential for negatively impacting intra- or postoperative course.
    2. Conditions that limit compliance with rehabilitation program.
    3. Any condition that has potential for significantly limiting patient's ability to assess postoperative ankle function.
    4. Any condition, psychiatric or otherwise, that would preclude informed consent/assent, consistent follow-up, or compliance with any aspect of the trial.
    5. Patient is currently abusing drugs or alcohol or, in the opinion of the Investigator, at high risk for poor compliance.
    6. Any result from screening blood work (including complete blood count, Prothrombin Time (PT)/Partial Thromboplastin Time (PTT)/INR, liver function, and creatinine) that exceeds 1.5x the upper limit of normal or is below 0.5x the lower limit of normal.

Ages: 17 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 309 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2030-07 (Estimated); Study Completion 2030-07 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline to Week 104 in the FAOS Pain and Function (SRA) subscale scores | Baseline to Week 104
  The FAOS is a 42-item, patient-reported outcome measure that assesses foot and ankle health in the past week. There are five FAOS subscales: Pain, Symptoms, Function (Daily Living), Function (SRA), and Foot and Ankle Related Quality of Life. The FAOS has been validated for a variety of foot and ankle conditions, including OLT. Responses to each question on the FAOS are recorded on a 5-point Likert scale. A normalized score out of 100 is calculated for each subscale, with 0 indicating extreme symptoms and 100 no symptoms.
  Selection of this composite primary endpoint is consistent with FDA guidance recommending selection of primary endpoints that evaluate changes in Pain and Function (SRA) subscale scores as they represent clinically meaningful outcomes for patients who receive products intended to repair or replace damaged cartilage in the knee.

SECONDARY OUTCOMES:
Percentage of subjects who respond to study treatment after 2 years, i.e., subjects who have ≥ 10-point improvement on both the FAOS Pain and Function (SRA) subscale scores from Baseline to Week 104. | Baseline to Week 104
  The FAOS is a 42-item, patient-reported outcome measure that assesses foot and ankle health in the past week. There are five FAOS subscales: Pain, Symptoms, Function (Daily Living), Function (SRA), and Foot and Ankle Related Quality of Life. The FAOS has been validated for a variety of foot and ankle conditions, including OLT. Responses to each question on the FAOS are recorded on a 5-point Likert scale. A normalized score out of 100 is calculated for each subscale, with 0 indicating extreme symptoms and 100 no symptoms.
Change from Baseline to Week 104 in the remaining FAOS subscales scores [Symptoms, Function (Daily Living) and Quality of Life] | Baseline to Week 104
  The FAOS is a 42-item, patient-reported outcome measure that assesses foot and ankle health in the past week. There are five FAOS subscales: Pain, Symptoms, Function (Daily Living), Function (SRA), and Foot and Ankle Related Quality of Life. The FAOS has been validated for a variety of foot and ankle conditions, including OLT. Responses to each question on the FAOS are recorded on a 5-point Likert scale. A normalized score out of 100 is calculated for each subscale, with 0 indicating extreme symptoms and 100 no symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathon Hopper BSc (Hons), MB ChB, FRCSEd, DIMC RCSEd., MBA, BSc (Hons), MB, Study Chair — Vericel Corporation
Locations (1):
- MedStar Georgetown University Hospital, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No